CLINICAL TRIAL: NCT01871584
Title: A Prospective, Single Center, Single-blinded, Randomized Study, of the Angel of Water™ for Colon Cleansing as Preparation for Colonoscopy
Brief Title: A Post Marketing Study of Angel of Water™ for Colon Cleansing as Preparation for Colonoscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: novoGI (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: Hydro-Prep, CLPR-200-0101
Record Dates: First submitted 2013-06-04; First posted 2013-06-06 (Estimated); Last update posted 2013-06-06 (Estimated); Status verified 2013-06

CONDITIONS: Colon Diseases
Keywords: A colon hydrotherapy system; Hydrocolonic preparation; Preparation for colonoscopy
MeSH Terms: conditions — Colonic Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hydrocolonic cleansing (Experimental): Subjects undergo colon cleansing by hydrotherapy with the study device
  Interventions: Device: Colon cleansing by hydrotherapy
- Standard preparation solution (Active Comparator): Subjects undergo colon cleansing by standard preparation solution
  Interventions: Device: Colon cleansing by hydrotherapy

INTERVENTIONS:
Device: Colon cleansing by hydrotherapy — The Angel of Water™ system will be used for hydrotherapy of the colon in adult subjects scheduled for elective colonoscopy.
  Other Names: The Angel of Water™, a colon hydrotherapy system.

SUMMARY:
The aim of this study is to demonstrate the efficacy of the hydrocolonic lavage method in order to prepare the colon prior to performing a colonoscopy, by comparison the hydrotherapy to standard preparation solution.

Hypothesis: Colon cleansing by hydrotherapy is as good as colon cleansing by standard preparation solution.

DETAILED DESCRIPTION:
Colonoscopy is the current standard method for evaluation of the colon. It has an indispensable place in the diagnosis and treatment of colon diseases. Diagnostic accuracy and therapeutic safety of colonoscopy depends on the quality of the colonic cleansing or preparation. Good preparation of the bowel is necessary prior to colonoscopy, to allow clear visualization of the bowel wall and any pathology within. The proposed study is a post-marketing study in which the study device, the Angel of Water system will be used for hydrotherapy of the colon in adult subjects scheduled for elective colonoscopy, instead of standard preparation solution. The effectiveness of the hydrotherapy in comparison to the standard preparation will be defined by evaluating colon cleanliness, subject's attitude and the duration of colonoscopy procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is >= 18 and ≤ 80 years old, referred to colonoscopy
2. Subject is able and agrees to sign the informed consent and follow the study requirements

Exclusion Criteria:

1. Myocardial infarction within the last 3 months
2. Symptomatic congestive heart failure
3. Established renal failure (serum creatinine > 2.0 mg/dL)
4. Previous abdominal surgery, colectomy, or recent colon or rectal surgery
5. Abdominal hernia
6. Partial or complete intestinal obstruction
7. Acute exacerbation of inflammatory bowel disease
8. Intestinal perforation
9. Fissures or fistula
10. Grade III or IV hemorrhoids
11. Carcinoma of the rectum
12. Distal rectal anastomosis
13. Cirrhosis
14. Hypokalemia
15. Pregnancy
16. Subject's weight > 400 lbs. /182 kg
17. Participation in another study that may affect the results of this study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2013-06; Primary Completion 2014-03 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Colon Cleanliness during colonoscopy according to Boston Bowel Preparation Scale (BBPS) | Per patient: the end of procedure; For study: approx. 10 months
  The primary study outcome is the Boston Bowel Preparation Scale (BBPS) score evaluating during colonoscopy. The BBPS is a valid scale for measuring bowel preparation as well as colonoscopy outcomes, as it reflects the colon's cleanliness during the inspection phase of the procedure.

SECONDARY OUTCOMES:
Subject's Attitude: rating the preparation procedure with respect to ease, convenience and comfort | Per patient: the end of procedure; For study: approx. 10 months
  Each subject will be asked to answer post cleansing questionnaire and a score will be calculated.

OTHER OUTCOMES:
Duration of colonoscopy examination | Per patient: the end of procedure; For study: approx. 10 months
  The duration of the colonoscopy procedure will be recorded for each subject. The duration is defined as the time from insertion into the rectum to the time when the colonoscopy is withdrawn across the anus.

CONTACTS AND LOCATIONS:
Overall Officials: Eran Choman, Study Director — novoGI
Locations (1):
- Department of Hepato-Gastroenterology, Nouvel Hopital Civil, Strasbourg, France